CLINICAL TRIAL: NCT00463047
Title: A Randomized, Double-Blind, Active-Controlled Crossover Study to Evaluate the Efficacy and Safety of Fentanyl Buccal Tablets Compared With Immediate-release Oxycodone for the Management of Breakthrough Pain in Opioid-Tolerant Patient With Chronic Pain
Brief Title: Efficacy and Safety of Fentanyl Buccal Tablets Compared With Oxycodone for the Management of Break Through Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: C25608/3055/BP/MN
Record Dates: First submitted 2007-02-08; First posted 2007-04-19 (Estimated); Results first posted 2010-12-14 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Pain
Keywords: Breakthrough pain; Opioid-tolerant; Chronic pain
MeSH Terms: conditions — Chronic Pain; Breakthrough Pain

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Fentanyl Buccal Tablets (FBT) (Experimental): This study includes a screening period, 2 open-label dose titration periods (in randomized order), and 2 double-blind treatment periods (in randomized order).
  Interventions: Drug: Fentanyl Buccal Tablets Compared With Immediate-Release Oxycodone
- Oxycodone (Active Comparator): This study includes a screening period, 2 open-label dose titration periods (in randomized order), and 2 double-blind treatment periods (in randomized order).
  Interventions: Drug: Fentanyl Buccal Tablets Compared With Immediate-Release Oxycodone

INTERVENTIONS:
Drug: Fentanyl Buccal Tablets Compared With Immediate-Release Oxycodone — Patients will be randomly assigned in a 1:1 ratio either to titrate immediate-release oxycodone first and to titrate FBT second, or to titrate FBT first and immediate-release oxycodone second, followed by 2 double-blind crossover treatment periods (in randomized order). For the double-blind treatment period of the study involving FBT administration, a patient is randomly assigned to receive FBT at the 200, 400, 600, or 800 mcg strength found to be successful during open-label titration. For the double-blind treatment period of the study to which a patient is randomly assigned to receive immediate-release oxycodone, the patient will receive immediate-release oxycodone at the strength (15, 30, 45, or 60 mg) found to be successful during open-label titration.

SUMMARY:
Evaluate the efficacy of treatment with Fentanyl Buccal Tablets (FBT) compared with immediate release oxycodone in alleviating breakthrough pain in opioid tolerant patients with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* The patient has chronic pain of at least 3 months duration associated with: diabetic peripheral neuropathy, postherpetic neuralgia, traumatic injury, complex regional pain syndrome, back pain, neck pain,fibromyalgia, chronic pancreatitis, osteoarthritis,or cancer.
* The patient is currently using 1 of the following: at least 60 mg of oral morphine/day, or at least 25 mcg of transdermal fentanyl/hour, or at least 30 mg of oxycodone/day, or at least 8 mg of hydromorphone/day, or an equianalgesic dose of another opioid/day as around-the-clock (ATC) therapy for at least 7 days before administration of the first dose of study drug
* The patient is willing to provide written informed consent to participate in this study.
* The patient is 18 through 80 years of age.
* Women must be surgically sterile, 2 years postmenopausal, or, if of childbearing potential, using a medically accepted method of birth control and agree to continued use of this method for the duration of the study.
* Any patient with cancer should have a life expectancy of at least 3 months.
* The patient reports an average Pain Intensity (PI) score, over the prior 24 hours, of 6 or less (0=no pain through 10=pain as bad as you can imagine) for their chronic pain.
* The patient experiences, on average, 1 to 4 breakthrough pain (BTP) episodes per day while taking ATC opioid therapy, and on average, the duration of each BTP episode is less than 4 hours.
* The patient currently uses opioid therapy for alleviation of BTP episodes, occurring at the location of the chronic pain, and achieves at least partial relief.
* The patient must be willing and able to successfully self-administer the study drug,comply with study restrictions, complete the electronic diary, and return to the clinic for scheduled study visits as specified in this protocol.

Exclusion Criteria:

* The patient has uncontrolled or rapidly escalating pain as determined by the investigator (i.e., the around-the-clock (ATC) therapy may be expected to change between the first and last treatments with study drug), or has pain uncontrolled by therapy that could adversely impact the safety of the patient or that could be compromised by treatment with study drug.
* The patient has a recent history (within 5 years) or current evidence of alcohol or other substance abuse.
* The patient has known or suspected hypersensitivities, allergies, or other contraindications to any ingredient in either study drug.
* The patient has cardiopulmonary disease that would, in the opinion of the investigator, significantly increase the risk of treatment with potent synthetic opioids.
* The patient has medical or psychiatric disease that, in the opinion of the investigator, would compromise collected data.
* The patient is expected to have surgery during the study that will impact the patient's chronic pain and/or BTP.
* The patient has had therapy before study drug treatment that, in the opinion of the investigator, could alter pain or response to pain medication.
* The patient is pregnant or lactating.
* The patient has participated in a previous study with FBT.
* The patient has participated in a study involving an investigational drug in the prior 30 days.
* The patient is currently using prescription FBT or immediate-release oxycodone for BTP and is unwilling to undergo re-titration.
* The patient has received a monoamine oxidase inhibitor (MAOI) within 14 days before the first treatment with study drug.
* The patient has any other medical condition or is receiving concomitant medication/therapy (eg, regional nerve block) that could, in the opinion of the investigator, compromise the patient's safety or compliance with the study protocol,or compromise collected data.
* The patient is involved in active litigation in regard to the chronic pain currently being treated.
* The patient has a positive urine drug screen (UDS) for an illicit drug or a medication not prescribed for him/her or which is not medically explainable.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2007-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (45):
- United States (45):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Birmingham Pain Center, Birmingham, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Desert Pain & Rehab Specialists/Redpoint Research, Phoenix, Arizona
  - Hope Research Institute, Phoenix, Arizona
  - Lovelace Scientific Resources, Inc., Beverly Hills, California
  - City of Hope National Medical Center, Duarte, California
  - Samaritan Center for Medical Research, Med. Group, Los Gatos, California
  - Advanced Diagnostic Pain Treatment Center, PC, New Haven, Connecticut
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Compass Research, Orlando, Florida
  - AvivoClin Clinical Services, Port Orange, Florida
  - Lovelace Scientific Resources, Inc., Sarasota, Florida
  - Clinical Research of Tampa Bay, Inc., Spring Hill, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - Center for Prospective Outcome Studies, Inc., Atlanta, Georgia
  - North Georgia Premier Research, Dawnsonville, Georgia
  - Taylor Research, LLC, Marietta, Georgia
  - DrugStudies America, Marietta, Georgia
  - Tristate Arthritis & Rheumatology Center, LLC, Evansville, Indiana
  - Rehabilitation Associates of Indiana, Indianapolis, Indiana
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - International Clinical Research Institute, Inc., Overland Park, Kansas
  - Kansas City Bone & Joint Clinic, Inc., Overland Park, Kansas
  - Willis-Knighton Pain Management Center, Shreveport, Louisiana
  - The Rehabilitation Team West, Baltimore, Maryland
  - Mid Atlantic Pain Medicine Center, Pikesville, Maryland
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - Metropolitan Hospital Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Raleigh Neurology Associate, Raleigh, North Carolina
  - Columbus Clinical Research, Columbus, Ohio
  - Allegheny Pain Management, Altoona, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Greenville Pharmaceutical, Greenville, South Carolina
  - Comprehensive Pain Specialists, PLLC, Hendersonville, Tennessee
  - Consultants in Pain Research, San Antonio, Texas
  - InVisions Consultants, LLC, San Antonio, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - The Center for Pain Relief, Charleston, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects 18 to 80 years of age with chronic pain for at least 3 months, were opioid tolerant, on around-the-clock opioid therapy, with 1-4 breakthrough pain episodes a day were recruited from 46 centers in the United States. First participant screened: June 2007. Last participant last visit: February 2009.
Pre-assignment Details: Prior to the double-blind treatment period, subjects participated in two titration periods to identify a "successful" and tolerated dose of Fentanyl Buccal Tablets (FBT) and immediate-release oxycodone. Subjects who did not titrate successfully were excluded from further participation in the study.
Groups:
- FBT First Immediate Release Oxycodone Second: Patients were randomized 1:1 to titrate Fentanyl Buccal Tablet (FBT) during the first titration period and then titrated immediate-release oxycodone during the second period or the reverse. Titration began with either 200 mcg FBT or 15 mg oxycodone taken as needed for breakthrough pain. If after 30 minutes pain relief was unsuccessful, a second dose could be taken. If more than one dose was required for at least 1 of 3 breakthrough pain episodes in one day, the next day the dose was increased in 200 mcg increments for FBT and 15 mg increments for oxycodone. The maximum allowable dose was 800 mcg for FBT (4 tablets) and 60 mg (4 capsules) for oxycodone. If a dose was not tolerated the dose was lowered to the previous tolerated dose. Titration completed when successful analgesia was achieved with a tolerated dose or maximum dose was reached. If unsuccessful at maximum dose subject was discontinued from proceeding further in the study. Subjects who successfully titrated were randomized.
- Immediate-Release Oxycodone First FBT Second: Patients were randomly assigned 1:1 to either titrate FBT during the first titration period and then titrated immediate-release oxycodone during the second period or the reverse. Titration began with either 200 mcg FBT or 15 mg oxycodone taken as needed for breakthrough pain. If after 30 minutes pain relief was unsuccessful, a second dose could be taken. If more than one dose was required for at least 1 of 3 breakthrough pain episodes in one day, the next day the dose was increased in 200 mcg increments for FBT and 15 mg increments for oxycodone. The maximum allowable dose was 800 mcg for FBT (4 tablets) and 60 mg (4 capsules) for oxycodone. If a dose was not tolerated the dose was lowered to the previous tolerated dose. Titration completed when successful analgesia was achieved with a tolerated dose or maximum dose was reached. If unsuccessful at maximum dose subject was discontinued from proceeding further in the study. Subjects who successfully titrated were randomized.
Period: Titration Period 1
Arm/Group | FBT First Immediate Release Oxycodone Second | Immediate-Release Oxycodone First FBT Second
Started | 160 (323 subjects entered study period but 3 discontinued before being randomized to treatment) | 160
Completed | 123 | 121
Not Completed | 37 | 39
Not completed — Adverse Event | 10 | 8
Not completed — Lack of Efficacy | 10 | 4
Not completed — Lost to Follow-up | 2 | 0
Not completed — Non-compliance with study medication | 3 | 5
Not completed — Protocol Violation | 5 | 5
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Non-compliance procedures | 4 | 10
Not completed — Other | 0 | 2
Period: Titration Period 2
Arm/Group | FBT First Immediate Release Oxycodone Second | Immediate-Release Oxycodone First FBT Second
Started | 123 | 121
Completed | 93 | 98
Not Completed | 30 | 23
Not completed — Adverse Event | 9 | 9
Not completed — Lack of Efficacy | 6 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 2 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Non-compliance study medication | 4 | 2
Not completed — Non-compliance procedures | 4 | 1
Not completed — Other | 3 | 2
Period: Double-Blind Treatment Period 1
Arm/Group | FBT First Immediate Release Oxycodone Second | Immediate-Release Oxycodone First FBT Second
Started | 96 (After completion of titration period subjects were re-randomized to these two treatment arms) | 94 (After completion of titration period subjects were re-randomized to these two treatment arms)
Completed | 93 | 90
Not Completed | 3 | 4
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 1 | 2
Not completed — Non-compliance with procedures | 1 | 0
Not completed — Other | 1 | 0
Period: Double-Blind Treatment Period 2
Arm/Group | FBT First Immediate Release Oxycodone Second | Immediate-Release Oxycodone First FBT Second
Started | 93 | 90
Completed | 92 | 88
Not Completed | 1 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Non-compliance with procedures | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Number of Patients: Fentanyl Buccal Tablets (FBT) and Immediate-Release Oxycodone crossover. The total number of patients (323) reflect the number that were enrolled to participate in the study prior to the first titration period. Three subjects withdrew before receiving any study drug so they are not listed as being assigned to either dosing arm in the titration studies, leaving only 320 subjects who were evenly divided between the two groups.
Arm/Group | Total Number of Patients
Number analyzed (Participants) | 323
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 323
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 50.2 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188
  Male | 135
Region of Enrollment [Number; unit: participants]
  United States | 323

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Difference (PID15) At 15 Minutes
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID15 is the difference between the PI scores from the episode baseline (immediately prior to study drug administration)and 15 minutes after the administration of the study drug. Least squared mean was from an analysis of variance (ANOVA) with treatment as randomized, phase, and sequence as fixed factors and patient as a random factor using compound symmetry.
Time Frame: Immediately pre-dose and fifteen minutes after administration of study drug
Population: Full Analysis Set defined as having at least one evaluable episode of breakthrough pain treated with FBT and at least one with oxycodone. An episode was evaluable if it had a valid pain intensity measurement immediately prior to drug administration. No imputation for missing breakthrough pain episodes, but LOCF was applied for missing PI scores.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Units Other Than Participants: breakthrough pain episodes
Groups:
- Fentanyl Buccal Tablets (FBT): FBT or matching placebo during the 2 double-blind treatment periods at doses of 200, 400, 600, and 800 mcg was self-administered by patients.
- Immediate-Release Oxycodone: Immediate-release oxycodone (or matching placebo) at doses of 15,30, 45, and 60 mg was self administered. The double-blind, treatment period used a 2 period crossover design in which the patient first managed 10 episodes with 1 of the 2 blinded study drugs (successful doses of immediate-release oxycodone or FBT) and then managed a subsequent 10 episodes with the other blinded study drug.
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Units on a scale | 0.82 (0.07) | 0.59 (0.07)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; The statistical hypothesis to be tested was:HO: µFBT = µOXY versus Ha: µFBT ≠ µoxy where µFBT and µOXY denote the mean PID15 for double-blind episodes for which patients use FBT and oxycodone (OXY), respectively. The primary variable was analyzed using a mixed effects ANOVA crossover model, with treatment as randomized (FBT or OXY), period, and treatment sequence (as randomized) as fixed factors and patient as a random factor, using compound symmetry for the variance-covariance matrix; Test type: Superiority or Other; p < 0.0001, Mixed effects ANOVA; Crossover analysis; Mean Difference (Final Values) = 0.23, 95% CI [0.18 to 0.29], Standard Error of Mean 0.07

2. Secondary Outcome: Pain Intensity Difference (PID 5) at 5 Minutes
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID5 is the difference between the PI score from the episode baseline (immediately prior to study drug administration) and 5 minutes after the administration of the study drug. Least squared mean was from an analysis of variance (ANOVA) with treatment as randomized, phase, and sequence as fixed factors and patient as a random factor using compound symmetry.
Time Frame: Immediately before and 5 minutes after study drug administration
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Units Other Than Participants: Episodes of breakthrough pain
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (Episodes of breakthrough pain) | 1764 | 1758
Units on a scale | 0.08 (0.03) | 0.05 (0.03)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; The statistical hypothesis to be tested was: HO: µFBT = µOXY versus Ha: µFBT ≠ µoxy where µFBT and µOXY denote the mean PID5 for double-blind episodes for which patients use FBT and OXY, respectively. The primary variable was analyzed using a mixed effects ANOVA crossover model, with treatment as randomized (FBT or OXY), period, and treatment sequence (as randomized) as fixed factors and patient as a random factor, using compound symmetry for the variance-covariance matrix; Test type: Superiority or Other; p = 0.0081, ANOVA — LS mean, SE of LS mean and p-value for treatment comparison are from ANOVA based on individual episodes with treatment as randomized, phase, and sequence as fixed factors and patient as random factor, using compound symmetry; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [0.01 to 0.05], Standard Error of Mean 0.03

3. Secondary Outcome: Pain Intensity Difference (PID 10) at 10 Minutes
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID10 is the difference between the PI score from the episode baseline (immediately prior to study drug administration) and 10 minutes after the administration of the study drug. Least squared mean was from an analysis of variance (ANOVA) with treatment as randomized, phase, and sequence as fixed factors and patient as a random factor using compound symmetry.
Time Frame: Immediately before and 10 minutes after administration of study drug
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Units on a scale | 0.30 (0.04) | 0.22 (0.04)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; The statistical hypothesis to be tested was: HO: µFBT = µOXY versus Ha: µFBT ≠ µoxy where µFBT and µOXY denote the mean PID10 for double-blind episodes for which patients use FBT and OXY, respectively. The primary variable was analyzed using a mixed effects ANOVA crossover model, with treatment as randomized (FBT or OXY), period, and treatment sequence (as randomized) as fixed factors and patient as a random factor, using compound symmetry for the variance-covariance matrix; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [0.05 to 0.13], Standard Error of Mean 0.04

4. Secondary Outcome: Pain Intensity Difference (PID 30) at 30 Minutes
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID30 is the difference between the PI score from the episode baseline (immediately prior to study drug administration) and 30 minutes after the administration of the study drug. Least squared mean was from an analysis of variance (ANOVA) with treatment as randomized, phase, and sequence as fixed factors and patient as a random factor using compound symmetry.
Time Frame: Immediately before and 10 minutes after study drug administration
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Units on a scale | 1.96 (0.09) | 1.58 (0.09)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.37, 95% CI [0.30 to 0.45], Standard Error of Mean 0.09

5. Secondary Outcome: Pain Intensity Difference (PID 45) at 45 Minutes
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID45 is the difference between the PI score from the episode baseline (immediately prior to study drug administration) and 45 minutes after the administration of the study drug. Least squared mean was from an analysis of variance (ANOVA) with treatment as randomized, phase, and sequence as fixed factors and patient as a random factor using compound symmetry.
Time Frame: Immediately before and 45 minutes after study drug administration
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Units on a scale | 2.87 (0.12) | 2.59 (0.12)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; The statistical hypothesis to be tested was: HO: µFBT = µOXY versus Ha: µFBT ≠ µoxy where µFBT and µOXY denote the mean PID45 for double-blind episodes for which patients use FBT and OXY, respectively. The primary variable was analyzed using a mixed effects ANOVA crossover model, with treatment as randomized (FBT or OXY), period, and treatment sequence (as randomized) as fixed factors and patient as a random factor, using compound symmetry for the variance-covariance matrix; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [0.20 to 0.35], Standard Error of Mean 0.12

6. Secondary Outcome: Pain Intensity Difference (PID 60) at 60 Minutes
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID60 is the difference between the PI score from the episode baseline (immediately prior to study drug administration) and 60 minutes after the administration of the study drug. Least squared mean was from an analysis of variance (ANOVA) with treatment as randomized, phase, and sequence as fixed factors and patient as a random factor using compound symmetry.
Time Frame: Immediately before and 60 minutes after administration of study drug
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Units on a scale | 3.35 (0.13) | 3.19 (0.13)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; The statistical hypothesis to be tested was: HO: µFBT = µOXY versus Ha: µFBT ≠ µoxy where µFBT and µOXY denote the mean PID60 for double-blind episodes for which patients use FBT and OXY, respectively. The primary variable was analyzed using a mixed effects ANOVA crossover model, with treatment as randomized (FBT or OXY), period, and treatment sequence (as randomized) as fixed factors and patient as a random factor, using compound symmetry for the variance-covariance matrix; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [0.08 to 0.25], Standard Error of Mean 0.13

7. Secondary Outcome: Percentage Change in Pain Intensity Difference (% PID) at 5 Minutes Post-treatment
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID5 is the difference between the PI scores from the episode baseline (immediately prior to study drug administration)and 5 minutes after the administration of the study drug. The difference is calculated and assessed as a percentage of the baseline pain intensity score. The percentage is calculated as the PID at 5 minutes divided by the baseline PI score times 100.
Time Frame: Immediately before and 5 minutes after administration of study drug
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent change in units on a scale
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Percent change in units on a scale | 1.11 (0.45) | 0.73 (0.37)

8. Secondary Outcome: Percentage Change in Pain Intensity Difference (%PID) at 10 Minutes
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID10 is the difference between the PI scores from the episode baseline (immediately prior to study drug administration)and 10 minutes after the administration of the study drug. The difference is calculated and assessed as a percentage of the baseline pain intensity score. The percentage is calculated as the PID at 10 minutes divided by the baseline PI score times 100.
Time Frame: Immediately before and 10 minutes after study drug administration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percentage change in units on a scale
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Percentage change in units on a scale | 4.08 (0.76) | 3.16 (0.57)

9. Secondary Outcome: Percentage Change in Pain Intensity Difference (%PID) at 15 Minutes
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID15 is the difference between the PI scores from the episode baseline (immediately prior to study drug administration)and 15 minutes after the administration of the study drug. The difference is calculated and assessed as a percentage of the baseline pain intensity score. The percentage is calculated as the PID at 15 minutes divided by the baseline PI score times 100.
Time Frame: Immediately before and 15 minutes after administration of study drug
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent change in units on a scale
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Percent change in units on a scale | 11.40 (1.15) | 8.59 (0.94)

10. Secondary Outcome: Percentage Change in Pain Intensity Difference (%PID) at 30 Minutes
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID30 is the difference between the PI scores from the episode baseline (immediately prior to study drug administration)and 30 minutes after the administration of the study drug. The difference is calculated and assessed as a percentage of the baseline pain intensity score. The percentage is calculated as the PID at 30 minutes divided by the baseline PI score times 100.
Time Frame: Immediately before and 30 minutes after study drug administration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent change in units on a scale
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Percent change in units on a scale | 27.83 (1.50) | 23.06 (1.33)

11. Secondary Outcome: Percentage Change in Pain Intensity Difference (% PID) at 45 Minutes
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID45 is the difference between the PI scores from the episode baseline (immediately prior to study drug administration)and 45 minutes after the administration of the study drug. The difference is calculated and assessed as a percentage of the baseline pain intensity score. The percentage is calculated as the PID at 45 minutes divided by the baseline PI score times 100.
Time Frame: Immediately before and 45 minutes after study drug administration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent change in units on scale
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Percent change in units on scale | 40.94 (1.76) | 37.56 (1.57)

12. Secondary Outcome: Percentage Change in Pain Intensity Difference (%PID) at 60 Minutes
Description: Pain intensity (PI) scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine after each episode of breakthrough pain during the double-blind treatment period. The PID60 is the difference between the PI scores from the episode baseline (immediately prior to study drug administration)and 60 minutes after the administration of the study drug. The difference is calculated and assessed as a percentage of the baseline pain intensity score. The percentage is calculated as the PID at 60 minutes divided by the baseline PI score times 100.
Time Frame: Immediately before and 60 minutes after study drug administration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent change in units on a scale
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Percent change in units on a scale | 48.08 (1.85) | 46.16 (1.75)

13. Secondary Outcome: Sum of Pain Intensity Difference at 30 Minutes Post-treatment (SPID30)
Description: PI scores were assessed on an 11-point numerical rating scale from 0 = no pain to 10 = pain as bad as you can imagine. SPID30 were derived from PID values. The SPID30 scores during the double-blind treatment phase were calculated as the time- weighted sum of the PID scores from 5 through 30 minutes,after the administration of study drug. SPID30 = (⅓ x PID5) + (⅓ x PID10) + (⅓ x PID15) + PID30. Least squared mean was from an analysis of variance (ANOVA) with treatment as randomized, phase, and sequence as fixed factors and patient as a random factor using compound symmetry.
Time Frame: From 5 minutes after dosing through 30 minutes after dosing
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Units on a scale | 2.36 (0.13) | 1.87 (0.13)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 0.49, 95% CI [0.39 to 0.58], Standard Error of Mean 0.13

14. Secondary Outcome: Sum of Pain Intensity Difference at 60 Minutes Post-treatment (SPID60)
Description: PI scores were assessed on an 11-point numerical rating scale from 0=no pain to 10=pain as bad as you can imagine during the double-blind treatment period. The SPID60 was derived from PID values. The SPID60 scores during the double-blind treatment phase were calculated as the time- weighted sum of the PID scores from 5 through 60 minutes,after the administration of the study drug.
  SPID60 = SPID30 + PID45 + PID60. Least squared mean was from an analysis of variance (ANOVA) with treatment as randomized, phase, and sequence as fixed factors and patient as a random factor using compound symmetry.
Time Frame: From 5 minutes after dosing through 60 minutes after dosing
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Units on a scale | 8.58 (0.34) | 7.65 (0.34)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 0.93, 95% CI 2-sided [0.70 to 1.16], Standard Error of Mean 0.34

15. Secondary Outcome: Pain Relief (PR) Score at 5 Minutes
Description: The PR score 5 minutes after the administration of study drug during the double-blind treatment phase was recorded in the patient's diary. The PR scale is a 5-point categorical scale of 0-4 (0=none, 1=slight, 2=moderate, 3=a lot, 4=complete).
Time Frame: Five minutes after administration of study drug
Population: Full Analysis Set defined as having at least one evaluable episode of breakthrough pain treated with FBT and at least one with oxycodone. An episode was evaluable if it had a valid pain intensity measurement immediately prior to drug administration. No imputation for missing breakthrough pain episodes, but LOCF was applied for missing PR scores.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 178 | 178
Units on a scale | 0.10 (0.43) | 0.09 (0.40)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; Test type: Superiority or Other; p = 0.1966, Wilcoxon (Mann-Whitney); P-value for the treatment comparison is from a one-sample Wilcoxon signed rank test

16. Secondary Outcome: Pain Relief Score (PR) at 10 Minutes
Description: The PR score 10 minutes after the administration of study drug during the double-blind treatment phase was recorded in the patient's diary. The PR scale is a 5-point categorical scale of 0-4 (0=none, 1=slight, 2=moderate, 3=a lot, 4=complete).
Time Frame: 10 minutes after treatment with study drug
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 178 | 178
Units on a scale | 0.30 (0.57) | 0.25 (0.53)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; Test type: Superiority or Other; p = 0.0275, Wilcoxon (Mann-Whitney); P-value for the treatment comparison is from a one-sample Wilcoxon signed rank test

17. Secondary Outcome: Pain Relief Score (PR) at 15 Minutes
Description: The PR score 15 minutes after the administration of study drug during the double-blind treatment phase was recorded in the patient's diary. The PR scale is a 5-point categorical scale of 0-4 (0=none, 1=slight, 2=moderate, 3=a lot, 4=complete).
Time Frame: 15 minutes after treatment with study drug
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 178 | 178
Units on a scale | 0.69 (0.74) | 0.53 (0.67)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; Test type: Superiority or Other; p = 0.0001, Wilcoxon (Mann-Whitney); P-value for the treatment comparison is from a one-sample Wilcoxon signed rank test

18. Secondary Outcome: Pain Relief Score (PR) at 30 Minutes
Description: The PR score 30 minutes after the administration of study drug during the double-blind treatment phase was recorded in the patient's diary. The PR scale is a 5-point categorical scale of 0-4 (0=none, 1=slight, 2=moderate, 3=a lot, 4=complete).
Time Frame: 30 minutes after treatment with study drug
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 178 | 178
Units on a scale | 1.50 (0.83) | 1.23 (0.76)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); P-value for the treatment comparison is from a one-sample Wilcoxon signed rank test

19. Secondary Outcome: Pain Relief Score (PR) at 45 Minutes
Description: The PR score 45 minutes after the administration of study drug during the double-blind treatment phase was recorded in the patient's diary. The PR scale is a 5-point categorical scale of 0-4 (0=none, 1=slight, 2=moderate, 3=a lot, 4=complete).
Time Frame: 45 minutes after treatment with study drug
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 178 | 178
Units on a scale | 2.08 (0.80) | 1.89 (0.74)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; Test type: Superiority or Other; p = 0.0004, Wilcoxon (Mann-Whitney); P-value for the treatment comparison is from a one-sample Wilcoxon signed rank test

20. Secondary Outcome: Pain Relief Score (PR) at 60 Minutes
Description: The PR score 60 minutes after the administration of study drug during the double-blind treatment phase was recorded in the patient's diary. The PR scale is a 5-point categorical scale of 0-4 (0=none, 1=slight, 2=moderate, 3=a lot, 4=complete).
Time Frame: 60 minutes after treatment with study drug
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 178 | 178
Units on a scale | 2.38 (0.76) | 2.24 (0.75)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; Test type: Superiority or Other; p = 0.0074, Wilcoxon (Mann-Whitney); P-value for the treatment comparison is from a one-sample Wilcoxon signed rank test

21. Secondary Outcome: Total Pain Relief (TOTPAR60) at 60 Minutes
Description: The mean TOTPAR at 60 minutes will be calculated for each episode as the weighted sum of Pain Relief (PR) scores (5-point Likert scale, 0 = none to 4 = complete) at each assessment of PR (during the double-blind treatment period) until 60 minutes after study drug administration, as follows:
  TOTPAR60 =(⅓ x PR5)+ (⅓ x PR10) +(⅓ x PR15)+ PR30 + PR45 + PR60. Least squared mean was from an analysis of variance (ANOVA) with treatment as randomized, phase, and sequence as fixed factors and patient as a random factor using compound symmetry.
Time Frame: From 5 minutes to 60 minutes after dosing
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 178 | 178
Number analyzed (breakthrough pain episodes) | 1676 | 1687
Units on a scale | 6.32 (0.16) | 5.63 (0.16)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.69, 95% CI [0.55 to 0.83], Standard Error of Mean 0.16

22. Secondary Outcome: Percent Total Pain Relief at 60 Minutes Posttreatment (%TOTPAR)
Description: The PR score at set intervals after the administration of study drug during the double-blind treatment phase was recorded in the patient's diary. The PR scale is a 5-point categorical scale of 0-4 (0=none, 1=slight, 2=moderate, 3=a lot, 4=complete). The maximum TOTPAR score that could be achieved at 60 minutes is equal to 16; thus, %TOTPAR at 60 minutes is (TOTPAR60 /16) times 100.The % TOTPAR achieved 60 minutes after the administration of study drug was calculated during the double-blind treatment phase.
Time Frame: From 5 minutes through 60 minutes after study drug treatment
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percent change in units on a scale
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 178 | 178
Percent change in units on a scale | 39.48 (15.67) | 35.28 (14.27)

23. Secondary Outcome: Time to Any Pain Relief (APR) by Treatment, <= 5 Minutes
Description: Time to APR was measured by stopwatch and by scheduled questions at each time point up to 60 minutes after baseline during double-blind treatment period. Any pain relief was defined as any subjective reduction in pain severity, even if not meaningful to patient. For each category (<5, <10, <15, <30, <45, <60 minutes, No APR-rescue medication used, and No APR-no rescue medication used)the number of episodes for which the time to APR fell into that category was compared. Here the number of episodes in which APR was achieved in less than or equal to 5 minutes was compared.
Time Frame: From time was administered to 5 minutes after treatment
Population: Full Analysis Set defined by at least one episode of breakthrough pain treated with FBT and at least one with oxycodone. No imputation was done if subject never answered APR/MPR question. If responded only as no, remaining missing imputed as no. If at least 1 yes, remaining missing imputed as yes.
Measure: Number; unit: Number of episodes treated
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Number of episodes treated | 48 | 33
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; Analysis is based on a generalized estimating equation model with treatment as a fixed effect and patient as a random effect. A logit link function and compound symmetry working correlation were applied in this model; Test type: Superiority or Other; p = 0.3022, Generalized estimating equation; Odds Ratio (OR) = 1.5054, 95% CI 2-sided [0.7 to 3.3]

24. Secondary Outcome: Time to Any Pain Relief (APR) by Treatment, <=10 Minutes
Description: The time to APR was measured by stopwatch and scheduled questions at each time point up to 60 minutes after baseline during the double-blind treatment periods. Any pain relief was defined as any subjective reduction in pain severity, even if not meaningful to patient. For each category (<5, <10, <15, <30, <45, <60 minutes, No APR-rescue medication used, and No APR-no rescue medication used)the number of episodes for which the time to APR fell into that category was compared. Here the number of episodes in which APR was achieved in less than or equal to 10 minutes was compared.
Time Frame: From study drug treatment until 10 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Number of episodes treated
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Number of episodes treated | 286 | 215
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.0268, Generalized estimating equation; Odds Ratio (OR) = 1.4042, 95% CI 2-sided [1.0 to 1.9]

25. Secondary Outcome: Time to Any Pain Relief (APR) by Treatment, <=15 Minutes
Description: The time to APR was measured by stopwatch and scheduled questions at each time point up to 60 minutes after baseline during double-blind treatment periods. Any pain relief was defined as any subjective reduction in pain severity, even if not meaningful to patient. For each category (<5, <10, <15, <30, <45, <60 minutes, No APR-rescue medication used, and No APR-no rescue medication used)the number of episodes for which the time to APR fell into that category was compared. Here the number of episodes in which APR was achieved in less than or equal to 15 minutes was compared.
Time Frame: From study drug administration to 15 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Number of episodes treated
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Number of episodes treated | 687 | 540
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.0008, Generalized estimating equation; Odds Ratio (OR) = 1.4631, 95% CI 2-sided [1.2 to 1.8]

26. Secondary Outcome: Time to Any Pain Relief (APR) by Treatment, <=30 Minutes
Description: The time to APR was measured by stopwatch and scheduled questions at each time point up to 60 minutes after baseline during double-blind treatment periods. Any pain relief was defined as any subjective reduction in pain severity, even if not meaningful to patient. For each category (<5, <10, <15, <30, <45, <60 minutes, No APR-rescue medication used, and No APR-no rescue medication used)the number of episodes for which the time to APRfell into that category was compared. Here the number of episodes in which APR was achieved in less than or equal to 30 minutes was compared.
Time Frame: Time of study drug administration till 30 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Number of episodes treated
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Number of episodes treated | 1259 | 1157
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.0084, Generalized estimating equation; Odds Ratio (OR) = 1.3184, 95% CI 2-sided [1.1 to 1.6]

27. Secondary Outcome: Time to Any Pain Relief (APR) by Treatment, <=45 Minutes
Description: The time to APR was measured by stopwatch and scheduled questions at each time point up to 60 minutes after baseline during double-blind treatment periods. Any pain relief was defined as any subjective reduction in pain severity, even if not meaningful to patient. For each category (<5, <10, <15, <30, <45, <60 minutes, No APR-rescue medication used, and No APR-no rescue medication used)the number of episodes for which the time to APRfell into that category was compared. Here the number of episodes in which APR was achieved in less than or equal to 45 minutes was compared.
Time Frame: Time of study drug treatment until 45 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Number of episodes treated
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Number of episodes treated | 1499 | 1480
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.5283, Generalize estimating equation; Odds Ratio (OR) = 1.0788, 95% CI 2-sided [0.9 to 1.4]

28. Secondary Outcome: Time to Any Pain Relief (APR) by Treatment, <=60 Minutes
Description: The time to APR was measured by stopwatch and scheduled questions at each time point up to 60 minutes after baseline during double-blind treatment periods. Any pain relief was defined as any subjective reduction in pain severity, even if not meaningful to patient. For each category (<5, <10, <15, <30, <45, <60 minutes, No APR-rescue medication used, and No APR-no rescue medication used)the number of episodes for which the time to APRfell into that category was compared. Here the number of episodes in which APR was achieved in less than or equal to 60 minutes was compared.
Time Frame: Time of study drug treatment until 60 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Number of episodes treated
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Number of episodes treated | 1559 | 1565
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.7110, Generalized estimating equation; Odds Ratio (OR) = 0.9491, 95% CI 2-sided [0.7 to 1.3]

29. Secondary Outcome: Time to Meaningful Pain Relief (MPR) by Treatment, <= 5 Minutes
Description: Time to MPR was measured by stopwatch and by scheduled questions at each time point up to 60 minutes after baseline during the double-blind treatment period. Meaningful pain relief was defined as a subject reduction of pain intensity that the subject found to be meaningful (substantive). For each category (<5, <10, <15, <30, <45, <60 minutes, No MPR-rescue medication used, and No MPR-no rescue medication used)the number of episodes for which the time to meaningful pain relief fell into that category was compared.
Time Frame: From time study drug was taken until 5 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Number of episodes treated
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Number of episodes treated | 9 | 18
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.3288, Generalized estimating equation; Odds Ratio (OR) = 0.5355, 95% CI 2-sided [0.2 to 1.9]

30. Secondary Outcome: Time to Meaningful Pain Relief (MPR) by Treatment, <=10 Minutes
Description: The time to MPR was measured by stopwatch and scheduled questions at each time point up to 60 minutes after baseline during double-blind treatment periods. Meaningful pain relief was defined as a subject reduction of pain intensity that the subject found to be meaningful (substantive). For each category (<5, <10, <15, <30, <45, <60 min, No MPR-rescue medication used, and No MPR-no rescue medication used)the number of episodes for which the time to MPR fell into that category was compared. Here the number of episodes in which MPR was achieved in less than or equal to 10 minutes was compared.
Time Frame: Time of study drug treatment until 10 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Number of episodes treated
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Number of episodes treated | 92 | 83
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.5145, Generalized estimating equation; Odds Ratio (OR) = 1.1485, 95% CI 2-sided [0.8 to 1.7]

31. Secondary Outcome: Time to Meaningful Pain Relief (MPR) by Treatment, <=15 Minutes
Description: The time to MPR was measured by stopwatch and scheduled questions at each time point up to 60 minutes after baseline during double-blind treatment periods. Meaningful pain relief was defined as a subject reduction of pain intensity that the subject found to be meaningful (substantive). For each category (<5, <10, <15, <30, <45, <60 min, No MPR-rescue medication used, and No MPR-no rescue medication used)the number of episodes for which the time to MPR fell into that category was compared. Here the number of episodes in which MPR was achieved in less than or equal to 15 minutes was compared.
Time Frame: Time of study drug administration until 15 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Number of episodes treated
Units Other Than Participants: breakthrough episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough episodes) | 1764 | 1758
Number of episodes treated | 286 | 211
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.0191, Generalized estimating equation; Odds Ratio (OR) = 1.4481, 95% CI 2-sided [1.1 to 2.0]

32. Secondary Outcome: Time to Meaningful Pain Relief (MPR) by Treatment, <=30 Minutes
Description: The time to MPR was measured by stopwatch and scheduled questions at each time point up to 60 minutes after baseline during double-blind treatment periods. Meaningful pain relief was defined as a subject reduction of pain intensity that the subject found to be meaningful (substantive). For each category (<5, <10, <15, <30, <45, <60 min, No MPR-rescue medication used, and No MPR-no rescue medication used)the number of episodes for which the time to MPR fell into that category was compared. Here the number of episodes in which MPR was achieved in less than or equal to 30 minutes was compared.
Time Frame: Time of study drug administration until 30 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Number of episodes treated
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Number of episodes treated | 787 | 636
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.0006, Generalized estimating equation; Odds Ratio (OR) = 1.4396, 95% CI 2-sided [1.2 to 1.8]

33. Secondary Outcome: Time to Meaningful Pain Relief (MPR) by Treatment, <=45 Minutes
Description: The time to MPR was measured by stopwatch and scheduled questions at each time point up to 60 minutes after baseline during double-blind treatment periods. Meaningful pain relief was defined as a subject reduction of pain intensity that the subject found to be meaningful (substantive). For each category (<5, <10, <15, <30, <45, <60 min, No MPR-rescue medication used, and No MPR-no rescue medication used)the number of episodes for which the time to MPR fell into that category was compared. Here the number of episodes in which MPR was achieved in less than or equal to 45 minutes was compared.
Time Frame: From study drug administration until 45 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Number of episodes treated
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Number of episodes treated | 1179 | 1060
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.0044, Generalized estimating equation; Odds Ratio (OR) = 1.3426, 95% CI 2-sided [1.1 to 1.6]

34. Secondary Outcome: Time to Meaningful Pain Relief (MPR) by Treatment, <=60 Minutes
Description: The time to MPR was measured by stopwatch and scheduled questions at each time point up to 60 minutes after baseline during double-blind treatment periods. Meaningful pain relief was defined as a subject reduction of pain intensity that the subject found to be meaningful (substantive). For each category (<5, <10, <15, <30, <45, <60 min, No MPR-rescue medication used, and No MPR-no rescue medication used)the number of episodes for which the time to MPR fell into that category was compared. Here the number of episodes in which MPR was achieved in less than or equal to 60 minutes was compared.
Time Frame: Time of study drug administration until 60 minutes after treatment
Population: as for outcome 23
Measure: Number; unit: Number of episodes treated
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Number of episodes treated | 1359 | 1313
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.2184, Generalized estimating equation; Odds Ratio (OR) = 1.1448, 95% CI 2-sided [0.9 to 1.4]

35. Secondary Outcome: Standard Rescue Medication Usage
Description: Any use of standard rescue medication after the administration of study drug for relief of Breakthrough Pain (BTP) during the double-blind treatment phase was recorded in the patient's diary. The number of breakthrough pain episodes for which study drug treatment was administered and which required rescue medication use was recorded.
Time Frame: During the administration of study drug during the double blind treatment periods.
Population: as for outcome 15
Measure: Number; unit: Number of episodes treated
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Number of episodes treated | 144 | 131
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.5808, Generalized estimating equation; Odds Ratio (OR) = 0.9249, 95% CI 2-sided [0.7 to 1.2]

36. Secondary Outcome: Medication Performance Assessment 30 Minutes After-treatment
Description: The medication performance assessment assessed study drug performance on a 5-point categorical scale of 0-4 (0=poor, 1=fair,2=good, 3=very good, 4=excellent) 30 minutes after administration of study drug during the double-blind treatment periods and for the first 5 BTP episodes after each visit during the open-label extension period were recorded in the patient's paper diary. Patients were asked "How well did your study medication perform in controlling this breakthrough pain episode?" The number of episodes rated for each category were recorded.
Time Frame: 30 minutes post-treatment
Population: as for outcome 15
Measure: Number; unit: Number of episodes treated
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Number of episodes treated
  Excellent | 45 | 18
  Very good | 153 | 104
  Good | 533 | 343
  Fair | 450 | 566
  Poor | 334 | 489
  No response | 249 | 238
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; Analysis is based on a generalized estimating equation model with treatment as a fixed effect and patient as a random effect. A cumulative logit link function and independent working correlation were applied in this model. Treatment differences for each time point were measured across all categories of responses; Test type: Superiority or Other; p < 0.0001, Generalized estimating equation; Odds Ratio (OR) = 1.8908, 95% CI 2-sided [1.7 to 2.2]

37. Secondary Outcome: Medication Performance Assessment 60 Minutes After-treatment
Description: The medication performance assessment assessed study drug performance on a 5-point categorical scale of 0-4 (0=poor, 1=fair,2=good, 3=very good, 4=excellent) 60 minutes after administration of study drug during the double-blind treatment periods and for the first 5 BTP episodes after each visit during the open-label extension period were recorded in the patient's paper diary. Patients were asked "How well did your study medication perform in controlling this breakthrough pain episode?" The number of episodes rated for each category were recorded.
Time Frame: 60 minutes post-treatment
Population: as for outcome 15
Measure: Number; unit: Number of episodes treated
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Number analyzed (breakthrough pain episodes) | 1764 | 1758
Number of episodes treated
  Excellent | 158 | 101
  Very good | 562 | 424
  Good | 679 | 726
  Fair | 210 | 335
  Poor | 128 | 146
  No response | 27 | 26
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets (FBT) vs Immediate-Release Oxycodone; [analysis description as in outcome 36, analysis 1]; Test type: Superiority or Other; p < 0.0001, Generalized estimating equation; Odds Ratio (OR) = 1.5841, 95% CI 2-sided [1.4 to 1.8]

38. Secondary Outcome: Breakthrough Pain Preference Questionnaire
Description: The BTP preference questionnaire is a questionnaire used to measure patients' preference for FBT or immediate-release oxycodone for management of BTP. The question is used to determine a patient's preference between the study drugs given in the 2 double-blind treatment periods. The patient was asked to select 1 of the following: 1, a preference for study drug used in the 1st double-blind treatment period; 2, a preference for study drug used in the 2nd double-blind treatment period; or 3, no preference.
Time Frame: After completion of both double-blind treatment periods or early termination
Population: Double-blind safety analysis set: 190 subjects who received both study drugs in this crossover study completed the Breakthrough Pain Preference Questionnaire after completing treatment
Measure: Number; unit: Participants
Groups:
- Total: Includes all patients who participated in the double-blind treatment period and completed treatment.
Arm/Group | Total
Number analyzed (Participants) | 190
Participants
  Preferred Fentanyl Buccal Tablet (FBT) | 99
  Preferred Immediate-Release Oxycodone | 63
  No preference | 15
  Missing | 13

39. Secondary Outcome: Pain Flare Treatment Satisfaction (PFTS) Questionnaire - Question 21 at the End of the First Double-blind Treatment Period (Visit 5)
Description: The PFTS is used to measure patient's satisfaction with study drug. Although the full scale has 25 questions, the question that is most useful (and least redundant with prior scales) for assessing the efficacy of the study drug is Question 21 which states: Which medication would you prefer to use when treating your pain flares? The subject can choose either: Prior medication, Study medication, or No preference. The number of subjects in each treatment group at the end of the first double-blind treatment period (Visit 5) who responded to each option is presented.
Time Frame: The end of the first double-blind treatment period.
Population: Double-blind safety analysis set: 88 subjects who received FBT and 90 subjects who received Oxycodone in the first double-blind period
Measure: Number; unit: Participants
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 88 | 90
Participants
  Prior Medication | 15 | 22
  Study Medication | 61 | 50
  No Preference | 12 | 18

40. Secondary Outcome: Pain Flare Treatment Satisfaction (PFTS) Questionnaire - Question 21 at the End of the Second Double-blind Treatment Period (Visit 6)
Description: The PFTS is used to measure patient's satisfaction with study drug. Although the full scale has 25 questions, the question that is most useful (and least redundant with prior scales) for assessing the efficacy of the study drug is Question 21 which states: Which medication would you prefer to use when treating your pain flares? The subject can choose either: Prior medication, Study medication, or No preference. The number of subjects in each treatment group at the end of the second double-blind treatment period (Visit 6) who responded to each option is presented.
Time Frame: At the end of the second double-blind treatment period (Visit 6)
Population: Double-blind safety analysis set: 83 subjects who received FBT and 87 subjects who received Oxycodone in the second double-blind period
Measure: Number; unit: Participants
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 83 | 87
Participants
  Prior Medication | 10 | 19
  Study Medication | 63 | 59
  No Preference | 10 | 9

41. Secondary Outcome: Pain Flare Treatment Satisfaction (PFTS) Questionnaire - Question 21 at Endpoint (End of Second Double-blind Treatment Period or Last Observation After Start of Treatment Period)
Description: The PFTS is used to measure patient's satisfaction with study drug. Although the full scale has 25 questions, the question that is most useful (and least redundant with prior scales) for assessing the efficacy of the study drug is Question 21 which states: Which medication would you prefer to use when treating your pain flares? The subject can choose either: Prior medication, Study medication, or No preference. The number of subjects in each treatment group at the Endpoint (time of the last observation during the treatment period)who responded to each option is presented.
Time Frame: Endpoint (End of second double-blind treatment period or last observation after start of treatment period)
Population: Double-blind safety analysis set: 88 subjects who received FBT and 94 subjects who received Oxycodone at any time during the double-blind treatment period who completed the PFTS questionnaire
Measure: Number; unit: Participants
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Number analyzed (Participants) | 183 | 183
Participants
  Prior Medication | 11 | 19
  Study Medication | 66 | 63
  No Preference | 12 | 12

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the two titration periods and double-blind treatment periods. Each titration period was 7-10 days in length and each double-blind treatment period was 7-17 days. The average duration of treatment was 24.2 days.
Description: 323 subjects were enrolled, 3 discontinued before receiving any study drug. 320 were randomized to titrate either FBT or oxycodone in first titration period. 36 received only FBT and discontinued (leaving 284 who received oxycodone), 39 received only oxycodone and discontinued leaving 281 who received FBT).
Groups:
- Fentanyl Buccal Tablets (FBT): FBT or matching placebo during the 2 double-blind treatment periods at doses of 200, 400, 600, and 800 mcg was self-administered by patients. This group includes all subjects in this study who had taken at least one dose of FBT in the course of the study, including both titration periods and both double-blind treatment periods. 320 subjects were randomized to titrate either FBT or oxycodone. 39 subjects received only oxycodone before discontinuing leaving 281 who received FBT during the study. 36 subjects received only FBT before discontinuing, leaving only 284 who received oxycodone.
- Immediate-Release Oxycodone: Immediate-release oxycodone (or matching placebo) at doses of 15,30, 45, and 60 mg was self administered. The double-blind, treatment period used a 2 period crossover design in which the patient first managed 10 episodes with 1 of the 2 blinded study drugs (successful doses of immediate-release oxycodone or FBT) and then managed a subsequent 10 episodes with the other blinded study drug. This arm represents all subjects who had exposure to at least one dose of immediate-release oxycodone either during the titration periods or double-blind periods. 320 subjects were randomized to titrate either FBT or oxycodone. 39 subjects received only oxycodone before discontinuing leaving 281 who received FBT during the study. 36 subjects received only FBT before discontinuing, leaving only 284 who received oxycodone.
Arm/Group | Fentanyl Buccal Tablets (FBT) | Immediate-Release Oxycodone
Serious Adverse Events (participants affected / at risk) | 1/281 | 0/284
Other Adverse Events (participants affected / at risk) | 79/281 | 49/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fentanyl Buccal Tablets (FBT) (N=281) | Immediate-Release Oxycodone (N=284)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl Buccal Tablets (FBT) (N=281) | Immediate-Release Oxycodone (N=284)
Nausea (Gastrointestinal disorders) | 26 | 11
Diarrhea (Gastrointestinal disorders) | 6 | 3
Vomiting (Gastrointestinal disorders) | 4 | 3
Constipation (Gastrointestinal disorders) | 1 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 3
Stomach discomfort (Gastrointestinal disorders) | 3 | 0
Application site pain (General disorders) | 13 | 0
Application site ulcer (General disorders) | 11 | 0
Fatigue (General disorders) | 2 | 4
Application site erythema (General disorders) | 5 | 0
Nasopharyngitis (Infections and infestations) | 4 | 3
Fall (Injury, poisoning and procedural complications) | 2 | 3
Headache (Nervous system disorders) | 12 | 8
Dizziness (Nervous system disorders) | 9 | 2
Somnolence (Nervous system disorders) | 6 | 5
Sedation (Nervous system disorders) | 3 | 2
Euphoric mood (Psychiatric disorders) | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 1
Application site irritation (General disorders) | 8 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days